CLINICAL TRIAL: NCT01056835
Title: Effects of PGI2 Analogue Use on the Development of Chronic Allograft Nephropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jongwon Ha, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Beraprost-01
Record Dates: First submitted 2010-01-24; First posted 2010-01-26 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Allograft Nephropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- control (No Intervention)
  Interventions: Drug: prostaglandin I2 analogue

INTERVENTIONS:
Drug: prostaglandin I2 analogue

SUMMARY:
The purpose of this study is to evaluate the effect of Prostaglandin I2 analogue use on the development of chronic allograft nephropathy and changes in allograft function in prevalent renal transplant recipients

ELIGIBILITY:
Inclusion Criteria:

* prevalent renal transplant recipients 2 years after transplantation
* no history of acute rejection
* stable renal function

Exclusion Criteria:

* history of biopsy-proven chronic allograft nephropathy
* history of biopsy-proven CNI nephrotoxicity
* history of biopsy-proven or clinical acute rejection
* unstable trough level of CNI or extremely low level of CNI
* bleeding tendency(+)
* pregnancy or pregnant-willing
* anticoagulation(+)
* antiplatelet agent (+)
* significant comorbidity(+): Acute coronary syndrome, pneumonia

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-06; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
graft pathology, serum creatinine, creatinine clearance, eGFR | 1 year after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Jongwon Ha, MD, PhD, Principal Investigator — Seoul National University
Locations (1):
- Seoul National University Hospital, Seoul, South Korea